CLINICAL TRIAL: NCT06747871
Title: Targeting Reinforcement Mechanisms for Smoking Cessation Using Very Low Nicotine Content Cigarettes in Individuals With Opioid Use Disorder and Chronic Pain
Brief Title: Opioids, Low Nicotine Cigarettes, and Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00116478; 1R34DA060477-01A1 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Tobacco Use; Opioid Substitution Treatment
MeSH Terms: conditions — Chronic Pain; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very Low Nicotine Cigarette (VLNC) Group (Experimental): Participants in this condition will be provided with VLNCs and asked to switch to smoking only study cigarettes for 4 weeks.
  Interventions: Behavioral: Very Low Nicotine Cigarettes (VLNC)
- Normal Nicotine Cigarette (NNC) Group (Active Comparator): Participants in this condition will be provided with NNCs and asked to switch to smoking only study cigarettes for 4 weeks.
  Interventions: Behavioral: Normal Nicotine Cigarettes (NNC)

INTERVENTIONS:
Behavioral: Very Low Nicotine Cigarettes (VLNC) — Spectrum NRC 102/103 (nonmenthol/ menthol) cigarettes, which have a nicotine content of approximately 0.4 mg/g tobacco.
  Arms: Very Low Nicotine Cigarette (VLNC) Group
Behavioral: Normal Nicotine Cigarettes (NNC) — Spectrum NRC 600/601 (nonmenthol/ menthol) cigarettes, which have a nicotine content of approximately 15.8 mg/g tobacco.
  Arms: Normal Nicotine Cigarette (NNC) Group

SUMMARY:
The purpose of this study is to evaluate the effects of switching to very low nicotine content (VLNC) cigarettes versus normal nicotine content (NNC) cigarettes on craving, withdrawal, and pain among individuals with chronic pain who smoke cigarettes daily and are attending office-based buprenorphine treatment (OBBT).

ELIGIBILITY:
Inclusion Criteria:

* Aged 21+ years who smoke cigarettes daily
* Chronic non-cancer musculoskeletal pain secondary to structural changes (e.g., low back pain, osteoarthritis)
* Have received stable office-based buprenorphine treatment for opioid use disorder for at least 30 days
* Self-report smoking at least 10 cigarettes/day
* Expired breath carbon monoxide (CO) level >8 ppm
* Have a smartphone capable of running software for ecological momentary assessment
* Open to exploring the possibility of quitting smoking

Exclusion Criteria:

* Pain specifically due to cancer
* Other significant health problems
* Major surgery within the past 6 months or planned surgery within the timeframe of the study
* Current disability litigation
* Use of electronic cigarettes or other non-cigarette tobacco products > 9 of the past 30 days
* Current use of nicotine replacement therapy or other cessation treatment
* Current daily or near-daily cannabis use
* History of psychotic disorder
* Acute suicidality or current unstable psychiatric disorder
* Positive pregnancy test
* Actively seeking smoking cessation treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Nicotine Dependence as measured by the Fagerstrom Test of Cigarette Dependence (FTCD) | Baseline and weekly during study cigarette use (4 weeks)
  The FTCD has a total score of 0 to 10, where a greater score indicates a greater physical dependence on nicotine.
Cigarettes per Day | Baseline and weekly during study cigarette use (4 weeks)
  Average cigarettes smoked per day during the past week will be calculated using timeline follow-back methods
Pain as measured by the Brief Pain Inventory (BPI) | Baseline, during abstinence sessions, and at weekly visits during study cigarette use (4 weeks)
  The BPI has an averaged score of 0 to 10, where a greater score indicates greater pain.
Mechanical Hyperalgesia | Weekly visits 1 and 5 during study cigarette use (4 weeks), and during abstinence sessions
  Mechanical hyperalgesia is a condition that causes increased sensitivity to mechanical stimuli after an injury to the skin. Discriminability and response bias will be assessed using a computerized pressure algometer.
Smoking Withdrawal as measured by the Minnesota Withdrawal Scale (MNWS) | Baseline, during abstinence sessions, and at weekly visits during study cigarette use (4 weeks)
  The MNWS has a total score range of 0 to 68, where a higher score indicates greater symptoms of withdrawal.
Cigarette Craving as measured by the Questionnaire of Smoking Urges-Brief (QSU-B) | Baseline, during abstinence sessions, and at weekly visits during study cigarette use (4 weeks)
  The QSU-B has a total score range of 0 to 100, where a higher score indicates greater craving.
Cigarette Purchase Task - demand intensity | Weekly visits 1 and 5 during study cigarette use (4 weeks), and during abstinence sessions
  Outcomes for the cigarette purchase task will include demand intensity (i.e., consumption at $0) and Omax (i.e., max expenditure at any price point).
Cigarette Purchase Task - Omax | Weekly visits 1 and 5 during study cigarette use (4 weeks), and during abstinence sessions
  Outcomes for the cigarette purchase task will include demand intensity (i.e., consumption at $0) and Omax (i.e., max expenditure at any price point).
Pain-Smoking Associations as measured by Ecological Momentary Assessment (EMA) | Baseline, weeks 1 and 4 of study cigarette use
  EMA (also called experience sampling or daily diary method) involves repeated sampling of people's current experiences (e.g. pain) in real time in their natural environments.
Buprenorphine-smoking associations as measured by Ecological Momentary Assessment (EMA) - smoking frequency | Baseline, weeks 1 and 4 of study cigarette use
  Within-person variability in smoking frequency assessed via EMA before and after buprenorphine administration.
Buprenorphine-smoking associations as measured by Ecological Momentary Assessment (EMA) - craving | Baseline, weeks 1 and 4 of study cigarette use
  Within-person variability in smoking craving assessed via EMA before and after buprenorphine administration.
Opioid Withdrawal as measured by the Short Opioid Withdrawal Scale (SOWS) | Baseline, during abstinence sessions, and at weekly visits during study cigarette use (4 weeks)
  The SOWS consists of 16 symptoms rated in intensity by patients on a 5-point scale of intensity as follows: 0-not at all, 1-a little, 2-moderately, 3-quite a bit, 4-extremely. The total score ranges from 0 to 64, where a higher score indicates greater symptoms of withdrawal.

SECONDARY OUTCOMES:
Number of participants willing to Quit Smoking | post-intervention, after 24 hrs abstinence
  Decision (yes/no) to engage in the optional quit attempt
Smoking abstinence self-efficacy as measured by the Self-Efficacy Questionnaire (SEQ) | Weekly visits 1 and 5
  The SEQ has a total score range of 10 to 40, where a higher score indicates greater self-efficacy.
Pain and Smoking Inventory (PSI) | Weekly visits 1 and 5
  The PSI total score is computed by averaging scores across the nine items. Items are endorsed on a seven-point Likert scale anchored at 0 (not true at all), 3 (somewhat true), and 6 (extremely true). Scores range from 0 to 6, where higher scores indicate greater perceptions that pain and smoking are interrelated.
Barriers to Quitting Smoking in Substance Abuse Treatment (BSQ-SAT) | Weekly visits 1 and 5
  The BQS-SAT is an 11-item true-false instrument of perceived barriers to quitting smoking plus one open-ended item. The score can range from 0 to 4.86, where a higher score indicates a greater perceived barrier.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Sweitzer, PhD, Principal Investigator — Duke University
Locations (1):
- North Pavilion, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include demographic, interview and self-report data. The investigators will share de-identified individual-participant level (IPD) data. Appropriate measures will be used for data de-identification and sharing, and informed consent will reflect those plans.